CLINICAL TRIAL: NCT02384954
Title: A Phase 1/2 Study of N-803 in Patients With Relapse/Refractory Indolent B Cell Non-Hodgkin Lymphoma in Conjunction With Rituximab
Brief Title: QUILT-3.002: N-803 in Patients With Relapse/Refractory iNHL in Conjunction With Rituximab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in drug product development strategy.
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-02-14
Record Dates: First submitted 2015-02-19; First posted 2015-03-10 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Indolent B Cell Non-Hodgkin Lymphoma
Keywords: Lymphoma; indolent B Cell; non-Hodgkin Lymphoma; Cancer; Immunotherapy; Relapsed; Refractory; Rituximab; Interleukin-15; Absolute Lymphocyte Count; White Blood Cell; Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; anti-CD20
MeSH Terms: conditions — Recurrence; Lymphoma; Lymphoma, Non-Hodgkin; Neoplasms; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Phase 1 Cohort 1: N-803 - IV 1 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 2: N-803 - IV 3 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 3: N-803 - IV 6 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 4: N-803 - SQ 6 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 5: N-803 - SQ 10 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 6: N-803 - SQ 15 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 1 Cohort 7: N-803 - SQ 20 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803
- Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg (Experimental)
  Interventions: Biological: Rituximab; Biological: N-803

INTERVENTIONS:
Biological: Rituximab — Intravenous infusion 375 mg/m^2.
  Other Names: Rituxin
Biological: N-803 — Intravenous infusion for Phase 1 cohort 1, 2 and 3; subcutaneous injection for Phase 1 cohort 4, 5, 6 and 7. Phase 2 dosing was based off of the MTD determined in Phase 1.

SUMMARY:
This is a Phase I/II, open-label, multi-center, competitive enrollment and dose escalation study of N-803 in patients with relapse/refractory indolent B cell non-Hodgkin lymphoma in conjunction with rituximab.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability, identify the Maximum Tolerated Dose (MTD) or the Minimum Efficacious Dose (MED) and designate a dose level for Phase 2. Also characterize the immunogenicity, pharmacokinetic profile, and biomarker serum levels of N-803 in treated patients.

The effect of N-803 on the peripheral absolute lymphocyte counts and white blood cell counts, the number, phenotype and repertoire of peripheral blood T (total and subsets) and NK cells will be evaluated. In addition, a subset of patients will be evaluated for changes in lymph node immune composition. Anti-tumor responses and survival data will also be collected in this trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of iNHL (Follicular lymphoma grade 1, 2, 3a; marginal zone lymphoma; small lymphocytic lymphoma or lymphoplasmacytic lymphoma) after treatment with at least 1 or more prior rituximab-containing regimens.

  * Anti-CD20 mAb-refractory disease is defined as progressive disease while on rituximab (or another treatment of an anti-CD20 monoclonal antibody) or progression within 6 months of rituximab-containing (or another treatment of an anti-CD20 antibody-containing) therapy.
  * Anti-CD20 mAb-sensitive disease is defined by a response to a prior rituximab-containing (or another treatment of an anti-CD20 monoclonal antibody) regimen, and relapse more than 6 months from the last administration of rituximab-containing (or another treatment of an anti-CD20 antibody-containing) therapy.
* Measurable disease:

  * At least one lymph node group ≥ 1.5 cm in longest transverse dimension. Patients with cutaneous only disease may be enrolled if they have a clearly measurable skin lesion.
  * Relapsed or Refractory iNHL that has progressed during or following 1 or more prior systemic rituximab-containing (or another treatment of an anti-CD20 antibody-containing) regimens for lymphoma

PRIOR/CONCURRENT THERAPY:

* No anti-lymphoma treatments within 28 days before the start of study treatment.
* Must have recovered from side effects of prior treatments.

PATIENT CHARACTERISTICS:

Performance Status

• ECOG 0, 1, or 2

Renal Function • Glomerular Filtration Rate (GFR) > 40mL/min or Serum creatinine ≤ 1.5 X ULN

Bone Marrow Reserve

* Platelets ≥30,000/uL
* Hemoglobin ≥ 8g/dL
* Absolute Lymphocytes ≥800/uL
* ANC/AGC ≥750/uL

Hepatic Function

* Total bilirubin ≤ 2.0 X ULN (unless Gilbert's Syndrome or disease infiltration of liver is present)
* AST, ALT ≤ 3.0 X ULN, or ≤ 5.0 X ULN (if liver lymphoma is present)
* No positive Hep C serology or active Hep B infection

Cardiovascular

* No congestive heart failure < 6 months
* No unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias or severe cardiac dysfunction
* No history of uncontrollable supraventricular arrhythmias
* No NYHA Class > II CHF
* No marked baseline prolongation of QT/QTc interval

Pulmonary

• Normal clinical assessment of pulmonary function

Other

* Negative serum pregnancy test if female and of childbearing potential
* Women who are not pregnant or nursing
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No known autoimmune disease other than corrected hypothyroidism
* No known prior organ allograft or allogeneic transplantation
* Not HIV positive
* No active CNS involvement with lymphoma
* No psychiatric illness/social situation that would limit compliance
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* Must provide informed consent and HIPPA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations
* No active systemic infection requiring parenteral antibiotic therapy
* No disease requiring systemic immunosuppressive therapy (inhaled or topical steroids are allowed). Adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* No known histologic transformation from iNHL to DLBCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine Oncology, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Foltz JA, Hess BT, Bachanova V, Bartlett NL, Berrien-Elliott MM, McClain E, Becker-Hapak M, Foster M, Schappe T, Kahl B, Mehta-Shah N, Cashen AF, Marin ND, McDaniels K, Moreno C, Mosior M, Gao F, Griffith OL, Griffith M, Wagner JA, Epperla N, Rock AD, Lee J, Petti AA, Soon-Shiong P, Fehniger TA. Phase I Trial of N-803, an IL15 Receptor Agonist, with Rituximab in Patients with Indolent Non-Hodgkin Lymphoma. Clin Cancer Res. 2021 Jun 15;27(12):3339-3350. doi: 10.1158/1078-0432.CCR-20-4575. Epub 2021 Apr 8. PMID 33832946
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33832946/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
Period: Phase 1
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
Completed | 1 | 3 | 1 | 2 | 3 | 3 | 3 | 0 | 0
Not Completed | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Failure to meet continuation criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 9 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
  years
    Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 21
    Phase 1 | 58.0 (1.00) | 64.7 (7.37) | 69.3 (8.39) | 60.0 (4.58) | 65.0 (10.44) | 68.3 (10.21) | 62.0 (3.61) |  |  | 63.9 (7.28)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9 | 25
    Phase 2 |  |  |  |  |  |  |  | 59.5 (11.39) | 69.1 (12.54) | 63.0 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
  Participants
    Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 21
    Phase 1: Female | 2 | 2 | 0 | 0 | 2 | 2 | 3 |  |  | 11
    Phase 1: Male | 1 | 1 | 3 | 3 | 1 | 1 | 0 |  |  | 10
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9 | 25
    Phase 2: Female |  |  |  |  |  |  |  | 10 | 2 | 12
    Phase 2: Male |  |  |  |  |  |  |  | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
  Participants
    Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 21
    Phase 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1: Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Phase 1: White | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 0 | 0 | 20
    Phase 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9 | 25
    Phase 2: American Indian or Alaska Native |  |  |  |  |  |  |  | 0 | 0 | 0
    Phase 2: Asian |  |  |  |  |  |  |  | 0 | 2 | 2
    Phase 2: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  | 0 | 0 | 0
    Phase 2: Black or African American |  |  |  |  |  |  |  | 0 | 1 | 1
    Phase 2: White |  |  |  |  |  |  |  | 14 | 6 | 20
    Phase 2: More than one race |  |  |  |  |  |  |  | 1 | 0 | 1
    Phase 2: Unknown or Not Reported |  |  |  |  |  |  |  | 1 | 0 | 1
Patients with relapse/refractory indolent B cell non-Hodgkin lymphoma [Count of Participants; unit: Participants] — Population: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
  Participants
    Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 21
    Phase 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |  | 21
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9 | 25
    Phase 2 |  |  |  |  |  |  |  | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: MTD or MED of N-803: IV 1, 3, 6 μg/kg, SQ 6, 10, 15, 20 μg/kg
Description: Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced Dose Limiting Toxicity (DLT) and that is one level below a dose that was not tolerated. Minimal Efficacious Dose (MED) is defined as a dose level which produces an Absolute Lymphocyte Count (ALC) ≥25,000/μL sustained for 14 days or a total WBC ≥35,000/μL sustained for 14 days among 2/3 or 4/6 of patients. The elevated ALC cannot be attributed to circulating lymphoma cells. Dose levels for N-803 1, 3, 6 μg/kg IV, and 6, 10, 15, 20 μg/kg subcutaneous (SQ) were used to determine the MTD or MED.
Time Frame: 9 months
Measure: Number; unit: SQ μg/kg
Groups:
- Phase 1 Cohort 7: N-803 - SQ 20 μg/kg: Rituximab: Intravenous infusion 375 mg/m^2.
  N-803: Intravenous infusion for Phase 1 cohort 1, 2 and 3; subcutaneous injection for Phase 1 cohort 4, 5, 6 and 7. Phase 2 dosing was based off of the MTD determined in Phase 1.
Arm/Group | Phase 1 Cohort 7: N-803 - SQ 20 μg/kg
Number analyzed (Participants) | 21
SQ μg/kg | 20

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment Emergent Adverse Event is defined as any AE that begins or worsens in grade after the start of study treatment until 30 days after the last dose of study treatment or end of study period, whichever is later.
Time Frame: 30 days after last dose, up to 40 weeks
Population: 3 subjects from Phase 1 cohort 7 rolled over to the Phase 2 portion of the study. All other participants in Phase 2 only enrolled in the Phase 2 portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 16 | 9
Participants
  Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
  Phase 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |
  Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9
  Phase 2 |  |  |  |  |  |  |  | 16 | 9

3. Primary Outcome: Overall Response Rate
Description: For Phase 1 and 2, overall response rate (ORR) will be calculated as the ratio of the number of patients who demonstrated response (CR+PR) divided by the number of patients in the Evaluable population. Response and disease progression criteria were defined by the 2007 IHP response assessments for malignant lymphoma.
Time Frame: 60 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 15 | 9
percentage of subjects
  Phase 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
  Phase 1 | 33 [0.8 to 90.6] | 33 [0.8 to 90.6] | 67 [9.4 to 99.2] | 33 [0.8 to 90.6] | 67 [9.4 to 99.2] | 67 [9.4 to 99.2] | 100 [29.2 to 100] |  |
  Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 9
  Phase 2 |  |  |  |  |  |  |  | 80 [51.9 to 95.7] | 33 [7.5 to 70.1]

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were to be reported within 30 days of the last dose of study treatment, regardless of attribution, up to 40 weeks. All deaths were followed during the disease progression and survival follow-up period, up to 42 months.
Arm/Group | Phase 1 Cohort 1: N-803 - IV 1 ug/kg | Phase 1 Cohort 2: N-803 - IV 3 ug/kg | Phase 1 Cohort 3: N-803 - IV 6 ug/kg | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/3 | 0/3 | 0/3 | 1/3 | 3/16 | 2/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 16/16 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: N-803 - IV 1 ug/kg (N=3) | Phase 1 Cohort 2: N-803 - IV 3 ug/kg (N=3) | Phase 1 Cohort 3: N-803 - IV 6 ug/kg (N=3) | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg (N=3) | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg (N=3) | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg (N=3) | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg (N=3) | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg (N=16) | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg (N=9)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: N-803 - IV 1 ug/kg (N=3) | Phase 1 Cohort 2: N-803 - IV 3 ug/kg (N=3) | Phase 1 Cohort 3: N-803 - IV 6 ug/kg (N=3) | Phase 1 Cohort 4: N-803 - SQ 6 ug/kg (N=3) | Phase 1 Cohort 5: N-803 - SQ 10 ug/kg (N=3) | Phase 1 Cohort 6: N-803 - SQ 15 ug/kg (N=3) | Phase 1 Cohort 7: N-803 - SQ 20 ug/kg (N=3) | Phase 2 Cohort 1: Anti-CD20 mAb-sensitive N-803 - SQ 20 ug/kg (N=16) | Phase 2 Cohort 2: Anti-CD20 mAb-refractory N-803 - SQ 20 ug/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 2
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 0 | 1 | 1 | 4 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 12 | 6
Fatigue (General disorders) | 1 | 2 | 3 | 1 | 1 | 3 | 3 | 7 | 6
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 13 | 8
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 4 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 1 | 2 | 3 | 3 | 13 | 9
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biopsy skin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 2
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papilloma excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT02384954/Prot_SAP_000.pdf